CLINICAL TRIAL: NCT03726463
Title: Evaluation of Intima and Media Layer of Iliac and Renal Artery to Verify a Mechanism of Intracranial Aneurysm Development in Autosomal Dominant Polycystic Kidney Disease Patients
Brief Title: Evaluation of Iliac and Renal Artery for Mechanism of Intracranial Aneurysm in ADPKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung Shin, Associate Professor, Asan Medical Center
Other Study IDs: 2018-1210
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Kidney Transplant; Complications; Polycystic Kidney Diseases; Aneurysm, Brain
MeSH Terms: conditions — Polycystic Kidney Diseases; Intracranial Aneurysm | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — renal artery, iliac artery, serum, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- polycystic kidney disease: patients with polycystic kidney disease who receive kidney transplantation at Asan Medical Center
  Interventions: Procedure: Kidney transplantation

INTERVENTIONS:
Procedure: Kidney transplantation — Bilateral nephrectomy of polycystic kidneys are routinely performed during kidney transplantation in ADPKD patients

SUMMARY:
ADPKD is the most common form of hereditary kidney disease and is known to occur in 1 of 400 to 1000 population in the U.S. ADPKD consists of 2.8% of patients receiving kidney transplantation in our center. It is known that ADPKD is associated with vascular anomalies, including abdominal aneurysms, valvular anomalies and especially intracranial aneurysms. Intracranial aneurysms occur in 9~12% of the ADPKD population which is higher than 2~3% in the general population and is known to be associated with PKD1 or PKD2 heritage.

Until now, most of the studies regarding intracranial aneurysms in ADPKD are conducted in animal models, and there are only few cellular studies conducted from human samples. While performing kidney transplantation to ESRD ADPKD patients, arterial tissues from nephrectomy specimens can be obtained. The objective of this study is to investigate the mechanism of intracranial aneurysm in ADPKD patients by analyzing iliac and renal artery characteristics.

DETAILED DESCRIPTION:
ADPKD is associated with PKD1 gene on chromosome 16 and PKD2 gene on chromosome 4 and these gene respectively code polycystin 1 and polycystin 2. Currently the hypotheses for increased intracranial aneurysm rate in ADPKD patients is that mutation of polycystin is not only confined to nephron tissues but also in endothelial cells and vascular smooth muscle cells and results in mutation of vascular phenotype. Also recent studies show polycystin complex causes cystic changes through mutation in primary cilia in renal epithelium. Wild type endothelial cells respond to fluid shear stress by regulating levels of intracellular calcium and nitric oxide, however, PKD1 or PKD2 mutation in fetal aortic endothelial cells revealed loss of these responses.

During kidney transplantation, bilateral nephrectomies are routinely performed to ADPKD patients. In this study, blood, urine, iliac artery and renal artery tissues will be collected from ADPKD patients receiving kidney transplantation to analyze the arterial characteristic and gene mutation of ADPKD patients. The aim of this study is to evaluate mechanisms associated with intracranial aneurysm occurence in ADPKD patients by analyzing the genetic mutation and vascular deformities of these patients.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients from ages 18 to 80 receiving kidney transplantation at Asan Medical Center

Exclusion Criteria:

* those who refuse or are unable to provide consent form
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADPKD patients from ages 18 to 80 receiving kidney transplantation at Asan Medical Center, which consists of approximately 2.8% of kidney transplantation patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Intracranial aneurysm | through study completion, average of 2 years
  Occurrence of intracranial aneurysm

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iglesias CG, Torres VE, Offord KP, Holley KE, Beard CM, Kurland LT. Epidemiology of adult polycystic kidney disease, Olmsted County, Minnesota: 1935-1980. Am J Kidney Dis. 1983 May;2(6):630-9. doi: 10.1016/s0272-6386(83)80044-4. PMID 6846334
- [Background] Collins AJ, Foley RN, Chavers B, Gilbertson D, Herzog C, Johansen K, Kasiske B, Kutner N, Liu J, St Peter W, Guo H, Gustafson S, Heubner B, Lamb K, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Thompson B, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Daniels F, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers P, Agodoa L. 'United States Renal Data System 2011 Annual Data Report: Atlas of chronic kidney disease & end-stage renal disease in the United States. Am J Kidney Dis. 2012 Jan;59(1 Suppl 1):A7, e1-420. doi: 10.1053/j.ajkd.2011.11.015. No abstract available. PMID 22177944
- [Background] Torres VE, Harris PC, Pirson Y. Autosomal dominant polycystic kidney disease. Lancet. 2007 Apr 14;369(9569):1287-1301. doi: 10.1016/S0140-6736(07)60601-1. PMID 17434405
- [Background] Ecder T, Schrier RW. Cardiovascular abnormalities in autosomal-dominant polycystic kidney disease. Nat Rev Nephrol. 2009 Apr;5(4):221-8. doi: 10.1038/nrneph.2009.13. PMID 19322187